CLINICAL TRIAL: NCT04308044
Title: Clinical Assessment of Pain Processes in Pediatric Patients With Chronic Musculoskeletal Pain
Acronym: MSK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Catherine Ferland, Principle Investigator, Shriners Hospitals for Children
Other Study IDs: A09-M17-17B
Record Dates: First submitted 2020-03-09; First posted 2020-03-13 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain
Keywords: Conditioned Pain Modulation; Chronic Musculoskeletal Pain; Quantitative Sensory Testing; Pain Management
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 10ml whole blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic MSK Pain: Participants who have chronic musculoskeletal pain.The pain profile of the patient will be assessed, including biological sample analysis (blood), quantitative sensory testing, electroencephalogram (EEG), and psychological state via the completion of questionnaires by the patient.
- Healthy Control: Participants who do not have chronic musculoskeletal pain.The pain profile of the patient will be assessed, including biological sample analysis (blood), quantitative sensory testing, electroencephalogram (EEG), insole assessment (40 healthy control participants), and psychological state via the completion of questionnaires by the patient.

SUMMARY:
Musculoskeletal (MSK) pain is one of the most common types of pain among children and adolescents. Recurring episodes of MSK pain during childhood does not only impact physical and psychological aspects of daily life but may predispose children and adolescents to experience recurrent pain-related illnesses while in adulthood. Thus, effective early life pain management is critical in avoiding a cascade of ill adaptive behaviors. Close to 16,000 children are seen in the clinics of the Shriners Hospital for Children - Canada each year. In the clinic, questionnaires are the standardized clinical way to access the patient's history on pain experience and their perception of it. However, clinicians currently lack the tools to objectively examine pain processes. The ultimate goal of this project is to investigate pain assessment techniques that could be used to phenotype pediatric MSK pain by their endogenous central pain modulation efficacy to provide a more personalized approach to pain management.

DETAILED DESCRIPTION:
Enabling better pain management in children with musculoskeletal (MSK) pathologies by improving assessment techniques is a cornerstone of this research program.

This research project will elucidate the regulation of specific physiological mechanisms related to pain in children reporting presence of chronic MSK pain. As molecular events of pathophysiological processes are quantifiable, the investigators will test for associations between the expression of pain-related molecular markers in blood and the patient's experience of pain assessed with semi-objective sensory testing. The identification of specific alterations in the nociceptive process will provide a deeper understanding of a patient's pain perception alongside self-report or observers' report subjective measurements. Pain experience variability may originate in the lack of rigor in the clinical pain assessment tools. A personalized mechanism-based approach may be the key to better identify a patient's pain outcome and how this assessment could lead to personalized pain management. By testing temporal summation (TS), conditioned pain modulation (CPM), electroencephalography (EEG) patterns and balance in relation to biomarkers, the investigators will be able to determine the phenotype of the patients who presents higher risk of central sensitization related to increased hyperactivity and decreased endogenous inhibition. The ultimate goal is to use this information to offer the highest quality of pain control in children with MSK conditions.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10 and 18 years old
* Report of MSK pain lasting 3 months or longer, including orthopaedic diagnoses such as those involving the spine, knees, hips, ankles, shoulders.
* Ability to adequately understand and respond to outcome measures
* Female or male
* Any ethnic background

Exclusion Criteria:

* Inability of the child to speak English or French
* Pain due to an acute trauma occurring in the last 3 months (e.g. fracture)
* Diagnosed with developmental delay that would interfere with understanding questions being asked (autism, mental retardation)
* Children with major chronic medical conditions (ASA status III or higher)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients will be recruited from outpatient clinics at the Shriners Hospitals for Children - Canada. Healthy participants will be recruited through word of mouth and recruitment advertisements in local magazines and social media. In collaboration with the public relations department of the hospital, previously-edited videos demonstrating the rationale and safety of the QST procedures mixed with interviews of past subjects will also be shared to promote the project and minimize potential concerns regarding our clinical assessment of pain.
Sampling Method: Non-Probability Sample
Enrollment: 518 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Mechanical detection threshold (grams) as measured with von Frey filaments | Completed during study visit (5 minutes).
Dynamic mechanical allodynia (numerical pain intensity using Faces Pain Scale -Revised scores 0-10) as measured with a standardized brush (Somedic SENSELab - Brush-05) | Completed during study visit (5 minutes).
Vibration detection threshold (Hertz) as measured with a Rydel-Seiffer graded tuning fork (64 Hz) | Completed during study visit (5 minutes).
Temporal mechanical summation (numerical pain intensity using Faces Pain Scale -Revised scores 0-10) as measured with the Neuropen (Owen Mumford) with disposable Neurotips | Completed during study visit (15 minutes).
Pain pressure threshold (Newtons) as measured with an algometer. | Completed during study visit (5 minutes).
Conditioned pain modulation (CPM) efficiency, a physiological parameter calculated as the percentage difference between the average pain intensity (0-10) reported during a thermode (heat) test before and after a cold water submersion bath test. | Completed during study visit (20 minutes).
Electroencephalography (EEG) (μV) as measured with a 24-electrode wireless EEG headset (DSI-24, Wearable Sensing) | Completed during study visit (5 minutes).
Biochemical assessment and genomic analysis of blood sample (10ml), drawn by research nurse. | The blood samples will be analyzed within 1 year of the study visit.
  A molecular assessment of monoamines involved in the dopaminergic and adrenergic pain (pathways related to the endogenous pain inhibitory system (dopamine, serotonin, epinephrine,norepinephrine) will be performed.
  Genomics analyses will be done to analyze specific single-nucleotide polymorphisms (SNPs). This process involves amplification of specific DNA fragments by polymerase chain reaction (PCR) followed by analysis on an optical plate for specific genetic polymorphisms, to identify which patients carry such polymorphisms.
Insole assessment (N; N/cm2; mm/s; mm) as measured with Moticon© sensor insoles | Completed during study visit (5 minutes).
  Forty participants who agree to participate in the insole assessment will be asked to stand on sensory insoles for a duration of fifteen seconds to measure the forces, pressures and center of pressure in their feet. The measurement data obtained using the Moticon© insoles will be aggregated for analysis of plantar pressure distribution, which will be performed using the Moticon© software.
Total score on Neuropathic Pain Questionnaire (DN4) (0-10) assessing the probability of neuropathic pain (score greater than 4 indicates neuropathic pain). | Completed during study visit (5 minutes).
  2 domains (Interview (0-7) and Examination (0-3) of the Patient) Completed by MSK chronic pain participants.
Total Score of the Functional Disability Inquiry (0-60). Higher scores indicate greater activity limitations during the past 2 weeks. | Completed during study visit (5 minutes).
  Completed by MSK chronic pain participants.
Total Subscale Score of the Adolescent Pediatric Pain Tool (APPT), which evaluates the intensity, location, and quality (including affective, evaluative, sensory, and temporal) dimensions of pain. | Completed during study visit (5 minutes).
  The APPT provides five subscale scores: 1) the number of pain sites (alternatively, the number of pain segments) as a measure of pain location from marks on a body outline; 2) a pain intensity score measured by a 10-centimeter line known as the Word Graphic Rating Scale (WGRS) and anchored by words no pain, little, medium, large, worst possible pain; 3) the number of pain quality descriptors, which yields percent scores for the sensory, affective, evaluative subscales; 4) the number of temporal descriptors, which yields a percent temporal subscale; and (5) the percent of total pain quality and temporal descriptors as a total subscale.
  Completed by MSK chronic pain participants.
Global Score of the Pittsburgh Sleep Quality Index (0-21). Higher scores indicate a worse sleep quality (>5 indicates "poor sleeper"). | Completed during study visit (5 minutes).
  Completed by all participants
Total Anxiety Score and Total Internalizing Scale on the Revised Children Anxiety and Depression Scale (RCADS) (0-47) (t-score of 65 = borderline clinical threshold, t-score 70 = above clinical threshold) | Completed during study visit (5 minutes).
  The RCADS is intended to assess children's report of symptoms corresponding to selected DSM-IV anxiety disorders and depression. .
  Scale yields Total Anxiety Score (5 anxiety subscales: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder), which gives an overall index of anxiety levels, and Total Internalizing Scale (sum of all 6 subscales, including major depression subscale), which provides an estimate of the total level of internalising symptoms.
  Completed by all participants.
Total Score of the Pain Catastrophizing Scale (0-52). Higher scores indicate higher levels of pain-related anxiety. | Completed during study visit (5 minutes).
  Completed by all participants.
Score of Trait Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater trait anxiety. | Completed during study visit (5 minutes).
  Completed by healthy control participant only.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ferland, PhD, Principal Investigator — Shriners Hospitals for Children,Canada
Locations (1):
- Shriners Hospital for Children-Canada, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No